CLINICAL TRIAL: NCT06874205
Title: Assessment of 11C-JMJ-129 for Imaging PDE4D in Brain and Whole Body of Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10001777; 001777-M
Record Dates: First submitted 2025-03-12; First posted 2025-03-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Healthy
Keywords: 11C-JMJ-129; PET Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One-arm (Other): All subjects will receive the same tests.
  Interventions: Drug: 11C-JMJ-129

INTERVENTIONS:
Drug: 11C-JMJ-129 — Injected IV followed by PET scanning

SUMMARY:
Background:

PDE4D is a protein in the body that plays a role in thinking and depression. This protein may play a major role in disorders such as Alzheimer disease or major depressive disorder. To learn more about these disorders, researchers want to be able to detect levels of PDE4D in the brain. 11C-JMJ-129 is a new radiotracer (a radioactive substance that highlights parts of the body during imaging scans) that was developed to attach only to PDE4D.

Objective:

To test the new radiotracer 11C-JMJ-129 during imaging scans in healthy volunteers.

Eligibility:

Healthy people aged 18 years and older who had a screening assessment under protocol 01-M-0254.

Design:

Participants will have 2 to 4 clinic visits.

Participants will be screened. They will have a physical exam. They will have blood tests and a test of their heart function.

Participants will undergo 1 or more of these scans:

A positron emission tomography (PET) scan of the whole body. The radiotracer will be injected through a tube placed in a vein in the arm. Participants will lie on a table while a donut-shaped machine passes over them. Blood will be drawn from the arm during this scan.

A magnetic resonance imaging (MRI) scan of the brain. Participants will lie on a table that slides into a tube.

A PET scan of the brain. These participants will be injected with the radiotracer. They will lie on a table with their head in the scanner.

Participants will be called within 3 days after each PET scan for a check on their health.

DETAILED DESCRIPTION:
Study Description:

This study is intended to provide information on the novel 11C-JMJ-129 radioligand and its ability to localize and measure PDE4D in the brain and body of healthy individuals.

Objectives:

Primary Objective: To study the brain uptake of 11C-JMJ-129 and perform kinetic modeling of the 11C-JMJ-129 in healthy individuals.

Secondary Objectives: To study brain retest variability and reliability, biodistribution, and dosimetry of 11C-JMJ-129 in healthy volunteers.

Endpoint:

Primary Endpoint: For both objectives, the primary endpoint is receptor density measured as distribution volume (VT).

Secondary Endpoint: Radiation burden to organs of the body.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Aged 18 years or older.
* Participants must have undergone a screening assessment under protocol 01-M-0254, "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Participants."
* Healthy based on medical history, physical examination, and laboratory testing.
* Able to provide informed consent.
* Willing and able to complete all study procedures including MRI tests.
* Have had their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Agree to adhere to the lifestyle considerations

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen).
* Any current Axis I diagnosis.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* History of seizures, other than in childhood and related to fever.
* Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours, including claustrophobia and weight greater than the maximum for the scanner (500 lbs).
* HIV Infection.
* Pregnancy or breast feeding.
* Participants must not have substance use disorder or alcohol use disorder.
* Unable to travel to the NIH.
* Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2029-02-05 (Estimated)

PRIMARY OUTCOMES:
Total Volume of Distribution | 120 minutes
  Quantification of JMJ129

SECONDARY OUTCOMES:
Dosimetry, ICC, aTRV, and biodistribution. | 120 minutes
  Quantification of JMJ129

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be submitted to ClinicalTrials.gov
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol.
Access Criteria: BTRIS

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001777-M.html